CLINICAL TRIAL: NCT04835844
Title: RHYTHMIA vs CARTO in Redo Ablation Procedures for Atrial Fibrillation: MAP-AF Study
Brief Title: RHYTHMIA vs CARTO in Redo Ablation Procedures for Atrial Fibrillation
Acronym: MAP-AF
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB 20-461
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mapping with CARTO: CARTO (Biosense Webster) in conjunction with CONFIDENSE mapping module and PENTARRAY catheter
  Interventions: Device: CARTO
- Mapping with RHYTHMIA: RHYTHMIA (Boston Scientific) in conjunction with the 64-electrodes ORION mini-basket catheter.
  Interventions: Device: RHYTHMIA

INTERVENTIONS:
Device: CARTO — Redo-ablation of paroxysmal AF with high density mapping system, CARTO, in conjunction with CONFIDENSE mapping module and PENTARRAY catheter
  Groups: Mapping with CARTO
Device: RHYTHMIA — Redo-ablation of paroxysmal AF with high density mapping system, RHYTHMIA, in conjunction with the 64-electrodes ORION mini-basket catheter.
  Groups: Mapping with RHYTHMIA

SUMMARY:
The MAP-AF study will compare RHYTHMIA vs CARTO in redo ablation of paroxysmal AF with assessment of both acute procedural profiles and clinical outcomes.

DETAILED DESCRIPTION:
Pulmonary venous conduction recovery is found in most patients undergoing redo ablation procedures for atrial fibrillation (AF). Identifying gaps in prior ablation lines is essential to achieve successful outcomes. High density mapping systems have been proposed to allow the identification of such gaps with speed and accuracy.

The MAP-AF study will compare RHYTHMIA vs CARTO in redo ablation of paroxysmal AF with assessment of both acute procedural profiles and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-90 years of age) undergoing redo ablation procedures for paroxysmal AF regardless of the systems or energy sources used during the pre-study ablation procedure(s).
* Paroxysmal AF: defined as AF terminating within 7 days of onset either spontaneously or with electrical or medical cardioversion.

Exclusion Criteria:

* Persistent AF
* Prior cardiac surgery
* Patients with only AFL or AT as the documented recurrent arrhythmia after the pre-study AF ablation(s).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Electrophysiology clinic patients who are considered candidates for redo paroxysmal AF ablation.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
System is able to accurately identify gaps | At the time of procedure
  Incidence of accurate identification of gaps in prior ablation lines by the system

SECONDARY OUTCOMES:
Treatment success | Up to 12 months
  Freedom from AF recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hussein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States